CLINICAL TRIAL: NCT06378255
Title: Clinical Evaluation of Polycation-based New Dental Desensitizer on Dentin Hypersensitivity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Hospital of Stomatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKUSSNCT-23A04; PKUSSIRB-202393160 (Other: Ethics Committee of PKUSH of Stomatology); Z221100007422088 (Other Grant/Funding Number: The SFP for clinical CDTT in capital)
Record Dates: First submitted 2024-04-16; First posted 2024-04-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dentin Sensitivity
Keywords: Dentin Sensitivity; Tooth desensitizer
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polycation-based new dentinal desensitizer (Experimental): Use a cotton ball or brush to apply a small amount of desensitizing agent to the sensitive tooth surface for about 1 minute and wait for 2 minutes. Excess gel is then wiped off the surface.
  Interventions: Device: Polycation-based new dentinal desensitizer
- GLUMA desensitizer (Placebo Comparator): Use according to instructions
  Interventions: Device: GLUMA desensitizer

INTERVENTIONS:
Device: Polycation-based new dentinal desensitizer — Dental desensitization treatment
  Arms: Polycation-based new dentinal desensitizer
Device: GLUMA desensitizer — Dental desensitization treatment
  Arms: GLUMA desensitizer

SUMMARY:
Evaluate the safety and clinical efficacy of new dental desensitizers in the treatment of dentin sensitivity, including the relief of sensitivity symptoms and the duration of efficacy.

DETAILED DESCRIPTION:
This is a randomized, single-blind and controlled study to include 40 patients with dentin sensitivity. The study will be a randomized controlled trial with split mouth control, with two quadrants of the same patient as test and control groups, the test group being the group using the new desensitizer and the control group being the group with the clinically used desensitizer (Gruma desensitizer). Improvement in dentin sensitivity symptoms was the primary outcome indicator observed. Dentin sensitivity was assessed by evaluating the reduction in dentin sensitivity VAS scores at immediately, 1 month, 3 months, and 6 months points after the desensitization treatment, and by evaluating the subjects' self-reported relief of sensitivity. Safety was assessed by evaluating appliance defects and adverse events at the immediately,1-, 3-, and 6-months points after the desensitization treatment.

ELIGIBILITY:
Inclusion Criteria:

* Dentin Hypersensitivity, with Vas score≥4 points and the normal pulp viability
* dentin-sensitive tooth in at least 2 different quadrants of the mouth (neck enamel dentin exposure or maxillofacial abrasion within the middle layer of dentin).
* in good overall health
* participants informed consent.

Exclusion Criteria:

* gastroesophageal reflux
* Dental caries, wedge defects, crowns or large fillings.
* Received dentin sensitivity desensitization treatment or used desensitization mouthwash within 1 month.
* Received systematic periodontal therapy or periodontal surgery within 3 months, ongoing orthodontic treatment, and medical treatment, including long-term use of anti-inflammatory, analgesic, and psychotropic medications.
* Pregnancy or breastfeeding.
* Participated in other clinical trials in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of dentin sensitivity induced by probe pressure stimulation | At Baseline and 10 minutes, 1 month, 3 months, 6 months after desensitization treatment
  The severity of dentin sensitivity is assessed using visual analogue scale (VAS) with numbers 0-10 by participants after probe pressure stimulation. Beforehand, the participants were informed that the 10 cm VAS would be used to assess their pain sensitivity, with 0 indicating no pain and 10 indicating the worst pain. Lower scores on the VAS indicate lower sensitivity. Dentin sensitivity was considered to have improved if the visual pain scale (F-VAS) score decreased by 2 or more points from baseline.

SECONDARY OUTCOMES:
Improvement of dentin sensitivity induced by air temperature stimulation | At Baseline and 10 minutes, 1 month, 3 months, 6 months after desensitization treatment
  The severity of dentin sensitivity is assessed using visual analogue scale (VAS) with numbers 0-10 by participants after cold air stimulation. Beforehand, the participants were informed that the 10 cm VAS would be used to assess their pain sensitivity, with 0 indicating no pain and 10 indicating the worst pain. Lower scores on the VAS indicate lower sensitivity. Dentin sensitivity was considered to have improved if the visual pain scale (F-VAS) score decreased by 2 or more points from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No